CLINICAL TRIAL: NCT01602523
Title: Effect of Symbicort on Sleep Quality in Patients With Emphysema
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Temple University (Other)
Responsible Party: Principal Investigator, Samuel Krachman, Principal Investigator, Professor of Medicine, Temple University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13383
Record Dates: First submitted 2012-04-23; First posted 2012-05-21 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Emphysema; Poor Sleep Quality
Keywords: Emphysema; COPD; Sleep
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- budesonide/formoterol (Active Comparator): budesonide/formoterol 160/4.5 mcg (Symbicort)
  Interventions: Drug: Budesonide/formoterol
- Placebo (Placebo Comparator): Symbicort placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide/formoterol — Budesonide/formoterol Spray inhaler 160/4.5 mcg daily 28 days
  Other Names: Symbicort
  Arms: budesonide/formoterol
Drug: Placebo — Placebo inhaler once daily 28 days
  Arms: Placebo

SUMMARY:
This study will look at the effects of the drug Symbicort on sleep quality. Symbicort is an inhaled medication that contains 2 drugs. One is a medication that opens up the airways (formoterol). The other is a steroid to decrease airway inflammation (budesonide). Symbicort is not an experimental medication. It is approved by the Food and Drug Administration for use in patients with emphysema. Patients with severe emphysema commonly sleep poorly. The cause of poor sleep in these patients is unknown. Symbicort may improve sleep quality by opening the airways and reducing lung inflammation. It is not known for sure if these effects actually improve sleep and quality of life. It is hoped that this study will answer this question.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe emphysema (GOLD stages 2 and 3)

Exclusion Criteria:

* Use of supplemental oxygen,
* A recent COPD exacerbation within the past 4 weeks.
* A previous diagnosis of obstructive sleep apnea
* A known urinary outflow obstruction,
* Glaucoma
* History of an allergic reaction to one of the study medications.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-04 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the objective assessment of sleep quality. | 28 days
  Sleep quality will be assessed quantitatively by polysomnogram and include measurement of sleep efficiency (total sleep time/time in bed), total sleep time, and arousal index during the night. Subjective sleep quality and assessment of daytime function will be measured using the Pittsburgh sleep quality index (PSQI) and the Epworth Sleepiness scale (ESS), respectively.

SECONDARY OUTCOMES:
Secondary outcome includes assessment of nocturnal oxygenation. | 28 days
  Nocturnal oxygenation will be measured by pulse oximetry.
Secondary outcome is the subjective assessment of sleep quality. | 28 days
  Quality of life will be assessed by SF-36 and SGRQ-C scores.
Secondary outcome includes assessment respiratory mechanics/function. | 28 days
  Respiratory function will be assessed by spirometry performed before sleep onset and upon awakening.
Secondary outcome includes assessment of overall quality of life. | 28 days
  Quality of life will be assessed by SF(short form)-36 and SGRQ-C(ST George's Respiratory Questionnaire for Chronic Obstructive Pulmonary Disease patients)scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Temple Lung Center, Philadelphia, Pennsylvania, United States